CLINICAL TRIAL: NCT03912233
Title: A Phase 2, Randomized, Double-blind, Controlled Study to Evaluate the Safety and Efficacy of VX-121 Combination Therapy in Subjects Aged 18 Years and Older With Cystic Fibrosis
Brief Title: A Study to Evaluate the Safety and Efficacy of VX-121 Combination Therapy in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX18-121-101
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor; tezacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part 1: Placebo (Placebo Comparator): Participants received placebo matched to VX-121/TEZ/VX-561 triple combination (TC) for 4 weeks in the treatment period and placebo matched to TEZ/VX-561 for 18 days in the washout period.
  Interventions: Drug: Placebo
- Part 1: VX-121/TEZ/VX-561 TC - Low Dose (Experimental): Participants received VX-121 5 milligram (mg) once daily (qd)/TEZ 100 mg qd/VX-561 150 mg qd TC for 4 weeks in the treatment period and TEZ 100 mg qd/VX-561 150 mg qd for 18 days in the washout period
  Interventions: Drug: VX-121; Drug: TEZ; Drug: VX-561
- Part 1: VX-121/TEZ/VX-561 TC - Medium Dose (Experimental): Participants received VX-121 10 mg qd/TEZ 100 mg qd/VX-561 150 mg qd TC for 4 weeks in the treatment period and TEZ 100 mg qd/VX-561 150 mg qd for 18 days in the washout period.
  Interventions: Drug: VX-121; Drug: TEZ; Drug: VX-561
- Part 1: VX-121/TEZ/VX-561 TC - High Dose (Experimental): Participants received VX-121 20 mg qd/TEZ 100 mg qd/VX-561 150 mg qd TC for 4 weeks in the treatment period and TEZ 100 mg qd/VX-561 150 mg qd for 18 days in the washout period.
  Interventions: Drug: VX-121; Drug: TEZ; Drug: VX-561
- Part 2: TEZ/IVA (Active Comparator): Following run-in period with TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) for 4 weeks, participants received TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the treatment period and TEZ 100 mg/IVA 150 mg q12h for 4 weeks in the washout period.
  Interventions: Drug: TEZ/IVA; Drug: IVA
- Part 2: VX-121/TEZ/VX-561 TC - High Dose (Experimental): Following run-in period with TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks, participants received VX-121 20 mg qd/TEZ 100 mg qd/VX-561 150 mg qd TC for 4 weeks in the treatment period and TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the washout period.
  Interventions: Drug: VX-121; Drug: TEZ; Drug: VX-561

INTERVENTIONS:
Drug: VX-121 — Tablets for oral administration.
  Arms: Part 1: VX-121/TEZ/VX-561 TC - High Dose; Part 1: VX-121/TEZ/VX-561 TC - Low Dose; Part 1: VX-121/TEZ/VX-561 TC - Medium Dose; Part 2: VX-121/TEZ/VX-561 TC - High Dose
Drug: TEZ — TEZ tablet for oral administration.
  Other Names: VX-661; Tezacaftor
  Arms: Part 1: VX-121/TEZ/VX-561 TC - High Dose; Part 1: VX-121/TEZ/VX-561 TC - Low Dose; Part 1: VX-121/TEZ/VX-561 TC - Medium Dose; Part 2: VX-121/TEZ/VX-561 TC - High Dose
Drug: VX-561 — Tablets for oral administration.
  Other Names: CTP-656; Deutivacaftor (D-IVA)
  Arms: Part 1: VX-121/TEZ/VX-561 TC - High Dose; Part 1: VX-121/TEZ/VX-561 TC - Low Dose; Part 1: VX-121/TEZ/VX-561 TC - Medium Dose; Part 2: VX-121/TEZ/VX-561 TC - High Dose
Drug: TEZ/IVA — Fixed-dose combination tablets for oral administration.
  Other Names: VX-661/VX-770; Tezacaftor/Ivacaftor
  Arms: Part 2: TEZ/IVA
Drug: IVA — Tablets for oral administration.
  Other Names: VX-770; Ivacaftor
  Arms: Part 2: TEZ/IVA
Drug: Placebo — Placebos matched to VX-121, TEZ, and VX-561 for oral administration.
  Arms: Part 1: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of VX-121 combination therapy in subjects with cystic fibrosis (CF).

ELIGIBILITY:
Key Inclusion Criteria:

* Part 1: Heterozygous for F508del and an MF mutation (F/MF)
* Part 2: Homozygous for F508del (F/F)
* FEV1 value ≥40% and ≤90% of the predicted mean for age, sex, and height

Key Exclusion Criteria:

* History of clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* History of solid organ or hematological transplantation

Other protocol-defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (12):
  - Keck Medical Center of University of Southern California, Los Angeles, California
  - Kaiser Permanente, Oakland, California
  - University of Kentucky., Lexington, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Santiago Reyes, M.D., Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Germany (3):
  - Charite Paediatric Pulmonology Department, Berlin
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Pneumologisches Studienzentrum Muenchen-West, München
- Netherlands (5):
  - Academic Medical Center, Amsterdam
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Heidelberglaan
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague
- Hospital de Santa Maria, Lisbon, Portugal
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, The Royal Victoria Infirmary, Newcastle upon Tyne
  - All Wales Adult Cystic Fibrosis Centre, University Hospital Llandough, Penarth

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Uluer AZ, MacGregor G, Azevedo P, Indihar V, Keating C, Mall MA, McKone EF, Ramsey BW, Rowe SM, Rubenstein RC, Taylor-Cousar JL, Tullis E, Yonker LM, Chu C, Lam AP, Nair N, Sosnay PR, Tian S, Van Goor F, Viswanathan L, Waltz D, Wang LT, Xi Y, Billings J, Horsley A; VX18-121-101; VX18-561-101 Study Groups. Safety and efficacy of vanzacaftor-tezacaftor-deutivacaftor in adults with cystic fibrosis: randomised, double-blind, controlled, phase 2 trials. Lancet Respir Med. 2023 Jun;11(6):550-562. doi: 10.1016/S2213-2600(22)00504-5. Epub 2023 Feb 23. PMID 36842446

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three parts were planned for this study, only Parts 1 (participants heterozygous for F508del and a minimal function mutation [F/MF genotypes]) and 2 (participants homozygous for F508del [F/F genotypes]) were conducted. Part 3 was optional and not conducted at sponsor's discretion.
Pre-assignment Details: A total of 87 participants were enrolled in this study (58 participants in Part 1 and 29 participants in Part 2 run-in Period), 1 participant in Part 2 run-in period discontinued from the study and was not randomized in the treatment period. Therefore, results are presented for 86 participants in this study.
Groups:
- Part 1: Placebo: Participants received placebo matched to VX-121/tezacaftor (TEZ)/VX-561 triple combination (TC) for 4 weeks in the treatment period and placebo matched to TEZ/VX-561 for 18 days in the washout period.
- Part 2: TEZ/IVA: Following run-in period with TEZ 100 mg qd/ivacaftor (IVA)150 mg every 12 hours (q12h) for 4 weeks, participants received TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the treatment period and TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the washout period.
Period: Overall Study
Arm/Group | Part 1: Placebo | Part 1: VX-121/TEZ/VX-561 TC - Low Dose | Part 1: VX-121/TEZ/VX-561 TC - Medium Dose | Part 1: VX-121/TEZ/VX-561 TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-121/TEZ/VX-561 TC - High Dose
Started | 10 | 9 | 19 | 20 | 10 | 18
Completed | 8 | 9 | 19 | 20 | 3 | 6
Not Completed | 2 | 0 | 0 | 0 | 7 | 12
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Placebo: Participants received placebo matched to VX-121/TEZ/VX-561 TC for 4 weeks in the treatment period and placebo matched to TEZ/VX-561 for 18 days in the washout period.
- Part 1: VX-121/TEZ/VX-561 TC - Low Dose: Participants received VX-121 5 mg qd/TEZ 100 mg qd/VX-561 150 mg qd TC for 4 weeks in the treatment period and TEZ 100 mg qd/VX-561 150 mg qd for 18 days in the washout period.
- Part 2: TEZ/IVA: Following run-in period with TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks, participants received TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the treatment period and TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the washout period.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: VX-121/TEZ/VX-561 TC - Low Dose | Part 1: VX-121/TEZ/VX-561 TC - Medium Dose | Part 1: VX-121/TEZ/VX-561 TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-121/TEZ/VX-561 TC - High Dose | Total
Number analyzed (Participants) | 10 | 9 | 19 | 20 | 10 | 18 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19 | 20 | 10 | 18 | 86
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 9 | 2 | 7 | 27
  Male | 8 | 5 | 16 | 11 | 8 | 11 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 10 | 8 | 19 | 17 | 8 | 18 | 80
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 9 | 8 | 18 | 17 | 9 | 18 | 79
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 3 | 1 | 0 | 5
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) [Count of Participants; unit: Participants] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  Participants
    <40 percent | 1 | 1 | 1 | 0 | 1 | 2 | 6
    >=40 to <70 percent | 9 | 6 | 14 | 17 | 6 | 11 | 63
    >=70 to <=90 percent | 0 | 2 | 4 | 3 | 3 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 Through Safety Follow-up (up to Day 75 for Part 1 and up to Day 85 for Part 2)
Population: Safety set included all participants who received at least 1 dose of study drug in the treatment period.
Measure: Number; unit: participants
Arm/Group | Part 1: Placebo | Part 1: VX-121/TEZ/VX-561 TC - Low Dose | Part 1: VX-121/TEZ/VX-561 TC - Medium Dose | Part 1: VX-121/TEZ/VX-561 TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-121/TEZ/VX-561 TC - High Dose
Number analyzed (Participants) | 10 | 9 | 19 | 20 | 10 | 18
participants
  Participants With AEs | 9 | 8 | 16 | 20 | 8 | 16
  Participants With SAEs | 2 | 1 | 1 | 0 | 0 | 0

2. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Day 29
Population: Full analysis set (FAS) included all randomized participants who carry the intended cystic fibrosis transmembrane conductance regulator gene (CFTR) allele mutation(s) and received at least 1 dose of study drug in the treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Part 1: Placebo | Part 1: VX-121/TEZ/VX-561 TC - Low Dose | Part 1: VX-121/TEZ/VX-561 TC - Medium Dose | Part 1: VX-121/TEZ/VX-561 TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-121/TEZ/VX-561 TC - High Dose
Number analyzed (Participants) | 10 | 9 | 19 | 20 | 10 | 18
percentage points | 1.9 [-4.1 to 8.0] | 4.6 [-1.3 to 10.6] | 14.2 [10.0 to 18.4] | 9.8 [5.7 to 13.8] | -0.1 [-6.4 to 6.1] | 15.9 [11.3 to 20.6]

3. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl) Concentrations
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Day 29
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Part 1: Placebo | Part 1: VX-121/TEZ/VX-561 TC - Low Dose | Part 1: VX-121/TEZ/VX-561 TC - Medium Dose | Part 1: VX-121/TEZ/VX-561 TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-121/TEZ/VX-561 TC - High Dose
Number analyzed (Participants) | 10 | 9 | 19 | 20 | 10 | 18
millimole per liter (mmol/L) | 2.3 [-7.0 to 11.6] | -42.8 [-51.7 to -34.0] | -45.8 [-51.9 to -39.7] | -49.5 [-55.9 to -43.1] | -2.6 [-8.2 to 3.1] | -45.5 [-49.7 to -41.3]

4. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline at Day 29
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part 1: Placebo | Part 1: VX-121/TEZ/VX-561 TC - Low Dose | Part 1: VX-121/TEZ/VX-561 TC - Medium Dose | Part 1: VX-121/TEZ/VX-561 TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-121/TEZ/VX-561 TC - High Dose
Number analyzed (Participants) | 10 | 9 | 19 | 20 | 10 | 18
units on a scale | 3.3 [-10.1 to 16.6] | 17.6 [3.5 to 31.6] | 21.2 [11.9 to 30.6] | 29.8 [21.0 to 38.7] | -5.0 [-16.9 to 7.0] | 19.4 [10.5 to 28.3]

5. Secondary Outcome: Observed Pre-dose Plasma Concentration (Ctrough) of VX-121, TEZ and Its Metabolite (M1-TEZ) and, VX-561 and Its Metabolites (M1-VX-561 and M6-VX-561)
Time Frame: Pre-dose at Day 15 and Day 29
Population: Pharmacokinetic (PK) set included all participants who received at least 1 dose study drug in the treatment period and for whom the PK data are considered sufficient and interpretable. Participants who received VX-121/TEZ/VX-561 TC in Parts 1 or 2 were to be analyzed for Ctrough. Overall participants in Part 1 were assessed for Ctrough, therefore data are reported in single Part 1: TC combined arm. The "number analyzed" signifies participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part 1: VX-121/TEZ/VX-561 TC - Combined: Participants who either received VX-121 5 mg, 10 mg or 20 mg qd/TEZ 100 mg qd/VX-561 150 mg qd TC for 4 weeks in the treatment period and TEZ 100 mg qd/VX-561 150 mg qd for 18 days in the washout period.
Arm/Group | Part 1: VX-121/TEZ/VX-561 TC - Combined | Part 2: VX-121/TEZ/VX-561 TC - High Dose
Number analyzed (Participants) | 48 | 18
nanogram per milliliter (ng/mL)
  Day 15: VX-121 5 mg: number analyzed (Participants) | 8 | 0
  Day 15: VX-121 5 mg | 317 (119) |
  Day 29: VX-121 5 mg: number analyzed (Participants) | 7 | 0
  Day 29: VX-121 5 mg | 366 (130) |
  Day 15: VX-121 10 mg: number analyzed (Participants) | 18 | 0
  Day 15: VX-121 10 mg | 520 (214) |
  Day 29: VX-121 10 mg: number analyzed (Participants) | 14 | 0
  Day 29: VX-121 10 mg | 582 (342) |
  Day 15: VX-121 20 mg: number analyzed (Participants) | 20 | 17
  Day 15: VX-121 20 mg | 974 (500) | 1050 (414)
  Day 29: VX-121 20 mg: number analyzed (Participants) | 18 | 16
  Day 29: VX-121 20 mg | 1160 (592) | 1030 (371)
  Day 15: TEZ: number analyzed (Participants) | 46 | 17
  Day 15: TEZ | 1890 (925) | 1870 (675)
  Day 29: TEZ: number analyzed (Participants) | 46 | 16
  Day 29: TEZ | 1920 (994) | 2070 (1340)
  Day 15: M1-TEZ: number analyzed (Participants) | 46 | 17
  Day 15: M1-TEZ | 4500 (1290) | 4550 (1200)
  Day 29: M1-TEZ: number analyzed (Participants) | 46 | 16
  Day 29: M1-TEZ | 4640 (1730) | 4440 (1680)
  Day 15: VX-561: number analyzed (Participants) | 46 | 17
  Day 15: VX-561 | 475 (247) | 457 (264)
  Day 29: VX-561: number analyzed (Participants) | 46 | 16
  Day 29: VX-561 | 510 (285) | 434 (257)
  Day 15: M1-VX-561: number analyzed (Participants) | 46 | 17
  Day 15: M1-VX-561 | 311 (141) | 326 (175)
  Day 29: M1-VX-561: number analyzed (Participants) | 46 | 16
  Day 29: M1-VX-561 | 336 (173) | 316 (188)
  Day 15: M6-VX-561: number analyzed (Participants) | 46 | 17
  Day 15: M6-VX-561 | 148 (98.0) | 174 (128)
  Day 29: M6-VX-561: number analyzed (Participants) | 46 | 16
  Day 29: M6-VX-561 | 163 (128) | 159 (94.6)

ADVERSE EVENTS:
Time Frame: From Day 1 Through Safety Follow-up (up to Day 75 for Part 1 and up to Day 85 for Part 2)
Groups:
- Part 2: TEZ/IVA: Following run-in period with TEZ 100 mg/IVA 150 mg q12h for 4 weeks, participants received TEZ 100 mg/IVA 150 mg q12h for 4 weeks in the treatment period and TEZ 100 mg/IVA 150 mg q12h for 4 weeks in the washout period.
Arm/Group | Part 1: Placebo | Part 1: VX-121/TEZ/VX-561 TC - Low Dose | Part 1: VX-121/TEZ/VX-561 TC - Medium Dose | Part 1: VX-121/TEZ/VX-561 TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-121/TEZ/VX-561 TC - High Dose
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/19 | 0/20 | 0/10 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/9 | 1/19 | 0/20 | 0/10 | 0/18
Other Adverse Events (participants affected / at risk) | 9/10 | 8/9 | 16/19 | 20/20 | 8/10 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=10) | Part 1: VX-121/TEZ/VX-561 TC - Low Dose (N=9) | Part 1: VX-121/TEZ/VX-561 TC - Medium Dose (N=19) | Part 1: VX-121/TEZ/VX-561 TC - High Dose (N=20) | Part 2: TEZ/IVA (N=10) | Part 2: VX-121/TEZ/VX-561 TC - High Dose (N=18)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=10) | Part 1: VX-121/TEZ/VX-561 TC - Low Dose (N=9) | Part 1: VX-121/TEZ/VX-561 TC - Medium Dose (N=19) | Part 1: VX-121/TEZ/VX-561 TC - High Dose (N=20) | Part 2: TEZ/IVA (N=10) | Part 2: VX-121/TEZ/VX-561 TC - High Dose (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 5 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 3 | 0
Fatigue (General disorders) | 0 | 2 | 5 | 2 | 2 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 1 | 2 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 4 | 3 | 0 | 3 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 2 | 2 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Viral rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 3 | 1 | 0 | 2
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 4 | 6 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Somnambulism (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 5 | 9 | 7 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 2 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 2 | 0 | 3
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 3 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 3 | 4 | 3 | 5
Throat clearing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT03912233/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT03912233/SAP_001.pdf